CLINICAL TRIAL: NCT03122808
Title: Intrapartum Uterine Activity Monitoring and Partogram Characteristics: Can They Help Predict Foetuses With Poor Tolerance of Labour?
Brief Title: Uterine Activity in Moderate-Severe Neonatal Encephalopathy: A Case Control Study
Status: Completed | Type: Observational
Sponsor: The Rotunda Hospital (Other)
Responsible Party: Principal Investigator, Breda Hayes, Consultant Neonatologist, The Rotunda Hospital
Other Study IDs: REC-2015-009
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Neonatal Encephalopathy
Keywords: Tachysystole; Excessive Uterine Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonatal encephalopathy: The inclusion criteria will be:
  * Moderate or severe neonatal encephalopathy
  * Gestational age of 35+0 weeks or greater
  * Singleton pregnancy
  * Inborn
  The exclusion criteria will be:
  * Non-hypoxic-ischaemic aetiology or postnatal hypoxic-ischaemia
  * Major congenital abnormalities
  * Less than 15 minutes of digital CTG recording from labour available
  Interventions: Diagnostic Test: Uterine Activity Analysis; Diagnostic Test: Partogram Analysis
- Control: The inclusion criteria will be:
  * Gestational age of 35+0 weeks or greater
  * Singleton pregnancy
  * Inborn
  The exclusion criteria will be:
  * APGAR score of less than 5 at 1 minute or less than 7 at 5 or 10 minutes
  * Admission to the neonatal unit
  * Major congenital abnormalities
  * Less than 15 minutes of digital CTG recording from labour available
  Interventions: Diagnostic Test: Uterine Activity Analysis; Diagnostic Test: Partogram Analysis

INTERVENTIONS:
Diagnostic Test: Uterine Activity Analysis — Analysis of components of uterine activity; contraction rate, length of contraction, length of relaxation and other values based off these measurements.
Diagnostic Test: Partogram Analysis — Analysis of slope of partogram

SUMMARY:
Excessive uterine activity may be one of several aetiological factors that contribute to depressed neurological function in the newborn. During labour, uterine contractions can compress the fetal cranium at pressures high enough to impair cerebral perfusion. Contraction rates greater than 7 in 15 minutes are associated with an increased risk of neonatal encephalopathy.

The American Congress of Obstetricians and Gynecologists defines uterine tachysystole as more than 5 contractions in 10 minutes, averaged over a 30-minute window. By this definition, excessive uterine activity is common and, at best, a non-specific predictor of depressed neurological function in the newborn. There is a need for predictors of neonatal encephalopathy that are more specific and clinically applicable.

Contraction and relaxation duration are two measures that closely reflect the proposed role of excessive uterine activity in the pathogenesis of neonatal encephalopathy. Prolonged contractions with short relaxation periods result in progressive reductions in fetal cerebral oxygenation. Shorter uterine contraction periods are associated with an increased risk of low umbilical cord potential of hydrogen (pH) values.

Our primary aim is to measure parameters of uterine activity, for example relaxation and contraction duration, and determine their relationship with the risk of neonatal encephalopathy. We will also investigate how measures of uterine activity interact with other measures of labour and fetal well-being, including cervical dilation rates and fetal heart rate patterns. In babies with neonatal encephalopathy, we will investigate the relationship of uterine activity with electrophysiological, radiological and developmental outcomes.

We will perform a retrospective case-control study of babies born in the Rotunda hospital from 2005 until the present. The assessor of the Cardiotocograph (CTG) recordings will be blind to the disease status of the infants. For each recording, every uterine contraction and rest interval will be measured. Summary variables created from these measures will be used to compare the case and control groups. The primary variable will be mean rest interval duration.

DETAILED DESCRIPTION:
The advent of therapeutic hypothermia has improved outcomes for babies born with hypoxic-ischemic encephalopathy. However, the risk of death, seizures, cerebral palsy or intellectual impairment remains significant, especially among the most severely affected infants. Prevention remains a promising strategy to reduce the incidence of complications arising from hypoxic-ischaemic neonatal encephalopathy.

Excessive uterine activity may be one of several aetiological factors that contribute to depressed neurological function in the newborn. During labour, uterine contractions can compress the fetal cranium at pressures high enough to impair cerebral perfusion. Contraction rates greater than 7 in 15 minutes are associated with an increased risk of neonatal encephalopathy.

The American Congress of Obstetricians and Gynecologists defines uterine tachysystole as more than 5 contractions in 10 minutes, averaged over a 30-minute window. By this definition, excessive uterine activity is common and, at best, a non-specific predictor of depressed neurological function in the newborn. There is a need for predictors of neonatal encephalopathy that are more specific and clinically applicable.

Contraction and relaxation duration are two measures that closely reflect the proposed role of excessive uterine activity in the pathogenesis of neonatal encephalopathy. Prolonged contractions with short relaxation periods result in progressive reductions in fetal cerebral oxygenation. Shorter uterine contraction periods are associated with an increased risk of low umbilical cord pH values.

Our primary aim is to measure parameters of uterine activity, for example relaxation and contraction duration, and determine their relationship with the risk of neonatal encephalopathy. We will also investigate how measures of uterine activity interact with other measures of labour and fetal well-being, including cervical dilation rates and fetal heart rate patterns. In babies with neonatal encephalopathy, we will investigate the relationship of uterine activity with electrophysiological, radiological and developmental outcomes.

We will perform a retrospective case-control study of babies born in the Rotunda hospital from 2005 until the present. Cases and controls must be over 35 weeks gestational age and have at least 15 minutes of Cardiotocograph (CTG) recording from labour available for analysis. Cases will be babies with moderate or severe neonatal encephalopathy of apparent hypoxic-ischemic aetiology. Controls will be the first healthy babies born before and after the cases to satisfy the study criteria. Controls will be matched for parity.

The assessor of the CTG recordings will be blind to the disease status of the infants. For each recording, every uterine contraction and rest interval will be measured. Summary variables created from these measures will be used to compare the case and control groups. The primary variable will be mean rest interval duration.

For further detail please see the study protocol.

ELIGIBILITY:
Cases

The inclusion criteria will be:

* Moderate or severe neonatal encephalopathy
* Gestational age of 35+0 weeks or greater
* Singleton pregnancy
* Inborn

The exclusion criteria will be:

* Non-hypoxic-ischaemic aetiology or postnatal hypoxic-ischaemia
* Major congenital abnormalities
* Less than 15 minutes of digital CTG recording from labour available Controls

The inclusion criteria will be:

* Gestational age of 35+0 weeks or greater
* Singleton pregnancy
* Inborn

The exclusion criteria will be:

* APGAR score of less than 5 at 1 minute or less than 7 at 5 or 10 minutes
* Admission to the neonatal unit
* Major congenital abnormalities
* Less than 15 minutes of digital CTG recording from labour available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is babies born in the Rotunda hospital since 2005, when digital archiving of cardiotocographs began. The Rotunda Hospital is a level 3 maternity hospital located in Ireland with approximately 9,000 deliveries per year. The incidence of moderate or severe neonatal encephalopathy in the population is approximately one per 1000 births.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Rest interval duration | Whole CTG recording from start of labour to delivery
  Expressed as mean, maximum, 90th centile. Individual uterine activity measures will be analysed both as continuous and categorised variables and in terms of minutes elapsed above a certain threshold that is to be determined.

SECONDARY OUTCOMES:
Rest interval as a percentage of contraction-rest interval cycle | Whole CTG recording from start of labour to delivery
  Expressed as mean, maximum, 90th centile. Individual uterine activity measures will be analysed both as continuous and categorised variables and in terms of minutes elapsed above a certain threshold that is to be determined.

OTHER OUTCOMES:
Contraction rate | Whole CTG recording from start of labour to delivery
  Expressed as mean, maximum, 90th centile. Individual uterine activity measures will be analysed both as continuous and categorised variables and in terms of minutes elapsed above a certain threshold that is to be determined.
Contraction duration | Whole CTG recording from start of labour to delivery
  Expressed as mean, maximum, 90th centile. Individual uterine activity measures will be analysed both as continuous and categorised variables and in terms of minutes elapsed above a certain threshold that is to be determined.
Excessive Uterine Activity Score | Whole CTG recording from start of labour to delivery
  Composite score based on combined assessment of contraction rate, contraction duration and relaxation time.

CONTACTS AND LOCATIONS:
Overall Officials: Breda Hayes, MD, Principal Investigator — The Rotunda Hospital
Locations (1):
- The Rotunda Hospital, Dublin, Co. Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No